CLINICAL TRIAL: NCT01420796
Title: Effect of Oral Motor Exercises and Breathing Exercises for Dysphagia in Parkinson Disease: Randomized Clinical Trial
Brief Title: Swallowing and Breathing Exercises for Dysphagia in Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Bahia (Other)
Responsible Party: Principal Investigator, Natalie Argolo Pereira Ponte, PhD, Federal University of Bahia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 96/10
Record Dates: First submitted 2011-08-18; First posted 2011-08-22 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Parkinson Disease; Dysphagia
Keywords: Parkinson's disease; dysphagia; swallowing treatment
MeSH Terms: conditions — Parkinson Disease; Deglutition Disorders | interventions — Breathing Exercises; Deglutition

STUDY DESIGN:
Intervention Model Description: 3 arms were designed to evaluate the effect of swallowing and breathing exercises to dysphagia in PD patients. The groups were allocated randomly in A) swallowing exercises; b) Breathing exercises or C) Swallowing and breathing exercises
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Swallowing and breathing exercises (Experimental): This group will perform both swallowing and breathing exercises for five weeks.
  Interventions: Other: Swallowing and breathing exercises
- Swallowing exercises (Experimental): This exercises aim to increase strength and range of motion of mouth, larynx and pharynx structures. All patients will perform sustained vowel phonation of /a/, pushing plosive phonemes /pa/, /ta/, /ka/ in a forceful manner, suction of wet gauze, swallowing with tongue hold and modified supraglottic maneuver, in ten repetitions, ascending and descending gliding phonation of vowel /a/ and /u/, five repetitions of each vowel, and tongue rotation in oral vestibule, 3 series of 5 repetitions to each side.
  Interventions: Other: Swallowing exercise
- Breathing exercises (Experimental): Expiratory Muscle Training will be performed with Threshold® (Respironics HealthScan, Inc, Cedar Grove, Nova Iorque, EUA).
  Interventions: Other: Breathing Exercises

INTERVENTIONS:
Other: Swallowing exercise — Patients will perform oral motor exercises for swallowing muscles for five weeks, four days a week.
  This exercises aim to increase strength and range of motion of mouth, larynx and pharynx structures. All patients will make sustained vowel phonation of /a/, pushing plosive phonemes /pa/, /ta/, /ka/ in a forceful manner, suction of wet gauze, swallowing with tongue hold and modified supraglottic maneuver, in ten repetitions, ascending and descending gliding phonation of vowel /a/ and /u/, five repetitions of each vowel, and tongue rotation in oral vestibule, 3 series of 5 repetitions to each side.
  Arms: Swallowing exercises
Other: Breathing Exercises — Patients will perform expiratory muscle training. Initial load will be 30% of maximal expiratory pressure which will increase until 75%. This load will be keep until end of training. Patients will made the exercises for 30 minutes with three minutes of training and two of rest.
  Arms: Breathing exercises
Other: Swallowing and breathing exercises — For five weeks, patients will perform swallowing and breathing exercises that follow: expiratory muscle training and sustained vowel phonation of /a/, pushing plosive phonemes /pa/, /ta/, /ka/ in a forceful manner, suction of wet gauze, swallowing with tongue hold and modified supraglottic maneuver, in ten repetitions, ascending and descending gliding phonation of vowel /a/ and /u/, five repetitions of each vowel, and tongue rotation in oral vestibule, 3 series of 5 repetitions to each side.
  Arms: Swallowing and breathing exercises

SUMMARY:
Parkinson's disease (PD) is a chronic, degenerative disease described by motors and non-motors symptoms. Changes in swallowing and respiratory dynamics increase risk of tracheal aspiration largely responsible for increased morbidity and mortality in this population. Thus, interdisciplinary rehabilitation strategies can reduce the complications of dysphagia, with consequent improvement of the prognosis of individuals with PD. Objective: To determine the impact of combined oral motor exercises and breathing exercises on swallowing disorders in individuals with PD. Method: Clinical trial, randomized and blinded for the examinator. For all subjects will be given the stage of PD and applied quality of life questionnaire. The swallowing complaints will be investigated through structured questionnaire and functional aspects of swallowing with videofluoroscopy. The Manovacuometry Spirometry will determine measures of respiratory function. The assessment of vocal and speech disorders will be done with perceptive, acoustic, aerodynamic and electroglottographic measures as well as analysis of intelligibility. Three groups of intervention will be defined: one of them doing oral motor exercises for swallowing, one doing breathing exercises and another must do this two interventions combined. Effect of intervention will be assessed through measures of swallowing, breathing, voice and speech. The groups will be compared, according to the principle of "intention to treat" by appropriate statistical tests, according to the distribution of the dependent variables.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease diagnosed following UKPDS Criteria
* Complaints and symptoms of dysphagia
* Dopaminergic treatment

Exclusion Criteria:

* Cranial trauma
* Severe heart disease
* Others neurologic disease
* Psychiatric diseases
* Therapy for swallowing or breathing in the last 3 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
Swallowing dynamics | five weeks
  Swallowing dynamics will be evaluated through videofluoroscopy of swallowing and electromyography.

SECONDARY OUTCOMES:
Vocal and speech measures | five weeks
  After recording a sample of speech, aerodynamics measures will be extracted by Aeroview Plus software and measures of test results electroglottography will be assessed on EG2 - PCX equipment.
Breathing measures | five weeks
  Spirometry will be made in KOKO® (software PDS Instrumentation, Inc., Louisville, Colorado, EUA), following American Thoracic Society protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Caline N. da Costa, Phd, Principal Investigator — DINEP/UFBA
Locations (1):
- Division of Neurology and Epidemiology, Salvador, Estado de Bahia, Brazil